CLINICAL TRIAL: NCT03016312
Title: A Phase III, Multicenter, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) in Combination With Enzalutamide Versus Enzalutamide Alone in Patients With Metastatic Castration-Resistant Prostate Cancer After Failure of an Androgen Synthesis Inhibitor and Failure of, Ineligibility for, or Refusal of a Taxane Regimen
Brief Title: A Study of Atezolizumab (Anti-PD-L1 Antibody) in Combination With Enzalutamide in Participants With Metastatic Castration-Resistant Prostrate Cancer (mCRPC) After Failure of an Androgen Synthesis Inhibitor And Failure of, Ineligibility For, or Refusal of a Taxane Regimen
Acronym: IMbassador250
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO39385; 2016-003092-22 (EudraCT Number)
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — atezolizumab; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Enzalutamide (Experimental): Participants will receive atezolizumab along with enzalutamide until investigator-assessed confirmed radiographic disease progression per PCWG3 criteria or unacceptable toxicity (up to approximately 42 months).
  Interventions: Drug: Atezolizumab; Drug: Enzalutamide
- Enzalutamide (Active Comparator): Participants will receive enzalutamide alone until investigator-assessed confirmed radiographic disease progression per PCWG3 criteria or unacceptable toxicity (up to approximately 42 months).
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1200 milligrams (mg), intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Other Names: Tecentriq®
  Arms: Atezolizumab + Enzalutamide
Drug: Enzalutamide — Enzalutamide capsules will be administered orally at a dose of 160 mg daily.
  Other Names: Xtandi®

SUMMARY:
This Phase III, multicenter, randomized, open-label study will evaluate the safety and efficacy of atezolizumab (anti-programmed death-ligand 1 [anti-PD-L1] antibody) in combination with enzalutamide compared with enzalutamide alone in participants with mCRPC after failure of an androgen synthesis inhibitor (e.g., abiraterone) and failure of, ineligibility for, or refusal of a taxane regimen. Participants will be randomized to one of the two treatment arms (atezolizumab in combination with enzalutamide, and enzalutamide alone) in a 1:1 ratio (experimental to control arm) in global randomized phase. Participants will receive treatment until investigator-assessed confirmed radiographic disease progression per Prostate Cancer Working Group 3 (PCWG3) criteria or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 3 months
* Histologically confirmed adenocarcinoma of the prostate
* Known castrate-resistant disease with serum testosterone level less than or equal to (</=) 50 nanograms per deciliter (ng/dL) with prior surgical castration or ongoing androgen deprivation for the duration of the study
* Progressive disease prior to screening by PSA or imaging per PCWG3 criteria during or following the direct prior line of therapy in the setting of medical or surgical castration
* One prior regimen/line of a taxane-containing regimen for mCRPC or refusal or ineligibility of a taxane-containing regimen
* Progression on a prior regimen/line of an androgen synthesis inhibitor for prostate cancer
* Availability of a representative tumor specimen from a site not previously irradiated that is suitable for determination of programmed death-ligand 1 (PD-L1) status via central testing
* Adequate hematologic and end organ function

Exclusion Criteria:

* Prior treatment with enzalutamide or any other newer hormonal androgen receptor inhibitor (e.g., apalutamide, ODM-201)
* Treatment with any approved anti-cancer therapy, including chemotherapy, immunotherapy, radiopharmaceutical or hormonal therapy (with the exception of abiraterone), within 4 weeks prior to initiation of study treatment
* Treatment with abiraterone within 2 weeks prior to study treatment
* Structurally unstable bone lesions suggesting impending fracture
* Known or suspected brain metastasis or active leptomeningeal disease
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study
* Active or history of autoimmune disease or immune deficiency
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Positive human immunodeficiency virus (HIV) test, active tuberculosis, active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Prior treatment with cluster of differentiation (CD)137 agonists or immune checkpoint blockade therapies, including anti Cytotoxic T Lymphocyte-Associated 4 (CTLA4), anti-programmed death 1 (PD-1), and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug, whichever is shorter, prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study
* History of seizure or any condition that may predispose to seizure within 12 months prior to study treatment, including history of unexplained loss of consciousness or transient ischemic attack

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (158):
- United States (39):
  - City of Hope Medical Grp Inc., Duarte, California
  - University of California San Diego, La Jolla, California
  - Kaiser Permanente San Diego - Los Angeles, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - University of Colorado; Division of Medical Oncology, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Stamford Hospital; BCC, MOHR, Stamford, Connecticut
  - Lynn Cancer Institute/Boca Raton Regional Hospital, Boca Raton, Florida
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Investigative Clin Rsch of IN, Indianapolis, Indiana
  - Associates in Oncology/Hematology P.C., Rockville, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute.., Detroit, Michigan
  - Nebraska Cancer Specialists; Oncology Hematology West, PC, Omaha, Nebraska
  - Urology Cancer Center & GU Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - MSKCC at Basking Ridge, Basking Ridge, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - James Cancer Hospital;Solove Research Institute, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute; Division of Medical Oncology, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Charleston Oncology, P .A, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology - Methodist Dallas Cancer Center, Dallas, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology-Tyler, Irving, Texas
  - Virginia Cancer Specialists - Alexandria, Alexandria, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Australia (6):
  - Eastern Health; Cancer Services, Box Hill, New South Wales
  - Concord Repatriation General Hospital; Concord Cancer Centre, Concord, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Royal Brisbane & Women's Hosp; Cancer Care Serv, Herston, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Monash Medical Centre; Oncology, Clayton, Victoria
- Austria (3):
  - LKH-UNIV. KLINIKUM GRAZ; Klinische Abteilung für Onkologie, Graz
  - Ordensklinikum Linz Elisabethinen; Abteilung für Urologie und Andrologie, Linz
  - Medizinische Universität Wien; Universitätsklinik für Urologie, Vienna
- Belgium (3):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - UZ Gent, Ghent
  - CHU Sart-Tilman, Liège
- Canada (8):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Kingston General Hospital, Kingston, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hopital Charles Lemoyne; Centre Integre de Lutte Contre Le Cancer de La Monteregie, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke - Hopital Fleurimont, Sherbrooke, Quebec
  - CHU de Québec - Université Laval - Hôtel-Dieu de Québec, Québec
- China (4):
  - Friendship Hospital, Capital Medical University, Beijing
  - Jiangsu Cancer Hospital, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Thomayerova nemocnice, Praha 4 - Krc
- Denmark (3):
  - Aalborg Universitetshospital; Onkologisk Afdeling, Aalborg
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- France (9):
  - Institut Sainte-Catherine; Oncologie, Avignon
  - Centre Francois Baclesse; Oncologie, Caen
  - Hopital Louis Pasteur; Medecine B, Colmar
  - Centre Oscar Lambret; Chir Cancerologie General, Lille
  - Clinique Chenieux; Oncology, Limoges
  - Hopital Saint Louis, Service D Oncologie Medicale, Paris
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Universitätsklinikum Freiburg; Chirurgische Klinik; Abteilung Urologie, Freiburg im Breisgau
  - Medizinische Hochschule Hannover; Klinik für Urologie und Onkologische Urologie, Hanover
  - Universitätsklinikum Münster, Klinik für Urologie und Kinderurologie, Münster
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
  - Urologisches Zentrum Euregio; Würselen, Urologische Praxis am Wasserturm, Würselen
- Greece (7):
  - Anticancer Hospital Ag Savas; 1St Dept of Internal Medicine, Athens
  - Alexandras Hospital; Dept. of Clin. Therapeutics, Athens Uni School of Medicine, Athens
  - Athens Medical Center; Dept. of Oncology, Athens
  - IASO General Hospital of Athens, Athens
  - Agioi Anargyroi Cancer Hospital; 2Nd Oncology Dept., Kifissia
  - University Hospital of Patras Medical Oncology, Pátrai
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Hungary (3):
  - Semmelwies University of Medicine; Urology Dept., Budapest
  - Orszagos Onkologiai Intezet; "C" Belgyógyászati-Onkológiai és Klinikai Farmakológiai Osztály, Budapest
  - Debreceni Egyetem Klinikai Kozpont ; Department of Oncology, Debrecen
- Italy (11):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - ISTITUTO NAZIONALE TUMORI IRCCS FONDAZIONE G. PASCALE; Dipartimento Uro-Ginecologico, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini; Oncologia Medica, Rome, Lazio
  - IRCCS AOU San Martino - IST; Oncologia Medica 1, Genoa, Liguria
  - A.O. Istituti Ospitalieri - Cremona; S.C. Oncologia, Cremona, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Cure Mediche, Milan, Lombardy
  - Ospedale Area Aretina Nord; U.O.C. Oncologia, Arezzo, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Prima, Padua, Veneto
- Japan (14):
  - Nagoya City University Hospital, Aichi
  - National Cancer Center East, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Yokohama City University Medical Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nara Medical University Hospital, Nara
  - Niigata University Medical & Dental Hospital, Niigata
  - Kansai Medical University Hospital, Osaka
  - Toranomon Hospital, Tokyo
  - The Jikei University Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
- Poland (8):
  - Woj. Wielospec. Centrum Onkologii i Traumatologii, ?ód?
  - Medical University of Bialystok; Oncology clinic, Bialystok
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - SPZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarawskiego, Opole
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Szpital Sw. Elzbiety - Mokotowskie Centrum Medyczne Sp. z o.o., Warsaw
  - Wojewodzki Szpital; Specjalistyczny ul., Wroclaw
- Russia (3):
  - Russian Scientific Center of Roentgenoradiology, Moscow, Moscow Oblast
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow, Moscow Oblast
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg, Sankt-Peterburg
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (13):
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Insititut Catala D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron; Oncology, Barcelona
  - Hospital Clínic i Provincial; Servicio de Oncología, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- Switzerland (2):
  - Inselspital Bern; Universitätsklinik für Medizinische Onkologie, Klinische Forschungseinheit, Bern
  - Kantonsspital St. Gallen; Onkologie/Hämatologie, Sankt Gallen
- Taiwan (4):
  - Taichung Veterans General Hospital; Division of Urology, Taichung
  - National Taiwan University Hospital, Department of Urology, Taipei
  - TAIPEI VETERANS GENERAL HOSPITAL, Urology, Taipei
  - Chang Gung Memorial Hospital-LinKou; Urology, Taoyuan District
- United Kingdom (6):
  - Royal Blackburn Hospital, Blackburn
  - Leicester Royal Infirmary, Leicester
  - Barts and the London NHS Trust., London
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital; Institute of Cancer Research, Sutton

REFERENCES:
- [Derived] Powles T, Yuen KC, Gillessen S, Kadel EE 3rd, Rathkopf D, Matsubara N, Drake CG, Fizazi K, Piulats JM, Wysocki PJ, Buchschacher GL Jr, Alekseev B, Mellado B, Karaszewska B, Doss JF, Rasuo G, Datye A, Mariathasan S, Williams P, Sweeney CJ. Atezolizumab with enzalutamide versus enzalutamide alone in metastatic castration-resistant prostate cancer: a randomized phase 3 trial. Nat Med. 2022 Jan;28(1):144-153. doi: 10.1038/s41591-021-01600-6. Epub 2022 Jan 10. PMID 35013615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 155 centres in 21 countries.
Pre-assignment Details: Total 759 participants were randomized.
Groups:
- Atezolizumab + Enzalutamide: Participants received atezolizumab along with enzalutamide until investigator-assessed confirmed radiographic disease progression per PCWG3 criteria or unacceptable toxicity.
- Enzalutamide: Participants received enzalutamide alone until investigator-assessed confirmed radiographic disease progression per PCWG3 criteria or unacceptable toxicity.
Period: Overall Study
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Started | 379 (participants randomized) | 380 (participants randomized)
Participants Received Treatment | 375 | 375
Completed | 17 | 10
Not Completed | 362 | 370
Not completed — discontinued before the treatment started | 0 | 1
Not completed — Withdrawal by Subject | 37 | 44
Not completed — Terminated by the Sponsor's decision | 100 | 126
Not completed — Physician Decision | 1 | 3
Not completed — Lost to Follow-up | 12 | 12
Not completed — Death | 210 | 184
Not completed — loss to contact | 1 | 0
Not completed — started a new cancer therapy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Total randomised participants 759.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide | Total
Number analyzed (Participants) | 379 | 380 | 759
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 90 | 187
  >=65 years | 282 | 290 | 572
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (8.3) | 70.6 (8.5) | 70.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 379 | 380 | 759
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 11 | 29
  Not Hispanic or Latino | 337 | 345 | 682
  Unknown or Not Reported | 24 | 24 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 71 | 65 | 136
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 7 | 14
  White | 279 | 287 | 566
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from randomization to death from any cause.
Time Frame: Baseline until death from any cause (up to approximately 42 months)
Population: The intent-to-treat (ITT) population is defined as all randomized participants regardless of whether the assigned study treatment was received. For efficacy analyses, participants were analyzed according to their randomized treatment assignment. Here, "Number Analyzed" refers to number of participants from whom data was collected and analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Months | 15.2 [14.0 to 17.0] | 16.6 [14.7 to 18.4]
Statistical Analysis 1: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Unstratified Analysis; Test type: Superiority; p = 0.0940, Log Rank; Hazard Ratio (HR) = 1.184, 95% CI 2-sided [0.971 to 1.445]
Statistical Analysis 2: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Stratified Analysis; Test type: Superiority; p = 0.2786, Log Rank; Hazard Ratio (HR) = 1.118, 95% CI 2-sided [0.913 to 1.370]

2. Secondary Outcome: Percentage of Participants Who Survived at Month 6 and 12
Description: OS (Overall Survival is defined as the time from randomization to death from any cause) probability at 6 and 12 months
Time Frame: Months 6, 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Percentage of Participants
  6 Months | 85.12 [81.45 to 88.78] | 85.32 [81.67 to 88.97]
  12 Months | 60.61 [55.52 to 65.71] | 64.65 [59.60 to 69.70]
Statistical Analysis 1: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Difference in Event Free Rate - 6 months; Test type: Superiority; p = 0.9391, z-test; Difference in Event Free Rate = -0.20, 95% CI 2-sided [-5.38 to 4.97]
Statistical Analysis 2: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Difference in Event Free Rate - 12 months; Test type: Superiority; p = 0.2706, z-test; Difference in Event Free Rate = -4.03, 95% CI 2-sided [-11.21 to 3.14]

3. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE)
Description: An SSE is defined as external beam radiation therapy to relieve skeletal symptoms (including initiation of radium-223 dichloride or other types of radionuclide therapy to treat symptoms of bone metastases), new symptomatic pathologic bone fracture, clinically apparent occurrence of spinal cord compression, or tumor related orthopedic surgical intervention.
Time Frame: Baseline up to end of study (up to approximately 42 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Months | 24.1 [24.1 to NA] — Due to censoring, the upper limit was not estimable. | 24.9 [24.9 to NA] — Due to censoring, the upper limit was not estimable.

4. Secondary Outcome: Radiographic Progression-Free Survival (rPFS), as Assessed by the Investigator and Adapted From the PCWG3 Criteria
Description: rPFS is defined as the time from randomization to the earliest occurrence of one of the following:
  * A participant is considered to have progressed by bone scan if: The first bone scan with ≥2 new lesions compared to baseline is observed < 12 weeks from randomization and is confirmed by a second bone scan taken ≥6 weeks later showing ≥2 additional new lesions (a total of ≥4 new lesions compared to baseline); the date of progression is the date of the first post-treatment scan, OR After the first post-treatment scan, ≥2 new lesions are observed relative to the first post-treatment scan, which is confirmed on a subsequent scan ≥6 weeks later; the date of progression is the date of the post-treatment scan when ≥2 new lesions were first documented.
  * Progression of soft tissue lesions, as defined per PCWG3 modified RECIST v1.1
  * Death from any cause
Time Frame: Baseline until disease progression or death from any cause (up to approximately 42 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Months | 4.2 [4.1 to 5.3] | 4.1 [3.7 to 4.5]
Statistical Analysis 1: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Unstratified Analysis; Test type: Superiority; p = 0.3157, Log Rank; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.775 to 1.086]
Statistical Analysis 2: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Stratified Analysis; Test type: Superiority; p = 0.2366, Log Rank; Hazard Ratio (HR) = 0.899, 95% CI 2-sided [0.754 to 1.072]

5. Secondary Outcome: Percentage of Participants Who Are Radiographic Progression-Free, as Assessed by the Investigator and Adapted From the PCWG3 Criteria
Description: as for outcome 4
Time Frame: Months 6, 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Percentage of Participants
  6 months | 41.84 [36.09 to 47.60] | 39.64 [33.86 to 45.42]
  12 months | 14.89 [10.74 to 19.05] | 13.45 [9.42 to 17.49]
Statistical Analysis 1: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Difference in Event Free Rate - 6 months; Test type: Superiority; p = 0.5959, z-test; Difference in Event Free Rate = 2.21, 95% CI 2-sided [-5.95 to 10.37]
Statistical Analysis 2: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Difference in Event Free Rate - 12 months; Test type: Superiority; p = 0.6262, z-test; Difference in Event Free Rate = 1.44, 95% CI 2-sided [-4.35 to 7.23]

6. Secondary Outcome: Percentage of Participants With Greater Than (>) 50 Percent (%) Decrease in Prostate-Specific Antigen (PSA) From Baseline
Description: PSA response rate, defined as a > 50% decrease in PSA from baseline that is confirmed after ≥ 3 weeks by a consecutive confirmatory PSA measurement
Time Frame: Baseline until disease progression (up to approximately 42 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Percentage of Participants | 25.9 [21.5 to 30.5] | 24.2 [20.0 to 28.7]
Statistical Analysis 1: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Test type: Superiority; Difference in 50% Decrease Response Rate = 1.6, 2% CI 2-sided [-4.5 to 7.8]; Odds Ratio: 1.1 95%CI: 0.8, 1.5

7. Secondary Outcome: Time to PSA Progression, Assessed as Per PCWG3 Criteria
Description: In participants with no PSA decline from baseline, PSA progression is defined as a ≥25% increase and an absolute increase of ≥2 ng/mL above the baseline value, ≥12 weeks after baseline. In participants with an initial PSA decline from baseline, PSA progression is defined as a ≥25% increase and an absolute increase of ≥2 ng/mL above the nadir value, which is confirmed by a consecutive second value obtained ≥3 weeks later.
Time Frame: Baseline until disease progression (up to approximately 42 months)
Population: The intent-to-treat (ITT) population is defined as all randomized participants regardless of whether the assigned study treatment was received. For efficacy analyses, participants were analyzed according to their randomized treatment assignment. Here, "Number Analyzed" refers to number of participants in the ITT population with measurable soft tissue lesions at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 379 | 380
Months | 2.8 [2.8 to 2.9] | 2.8 [2.8 to 2.9]
Statistical Analysis 1: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Unstratified Analysis; Test type: Superiority; p = 0.5359, Log Rank; Hazard Ratio (HR) = 1.055, 95% CI 2-sided [0.890 to 1.251]
Statistical Analysis 2: Comparison: Atezolizumab + Enzalutamide vs Enzalutamide; Stratified Analysis; Test type: Superiority; p = 0.6857, Log Rank; Hazard Ratio (HR) = 1.037, 95% CI 2-sided [0.869 to 1.238]

8. Secondary Outcome: Percentage of Participant With Objective Response, as Determined by the Investigator Through Use of PCWG3 Criteria
Description: Objective response rate in soft tissue lesions, defined as the percentage of participants with either a CR or PR on two consecutive occasions ≥ 6 weeks apart, as determined by the investigator through use of PCWG3 criteria
Time Frame: Baseline until disease progression or death from any cause (up to approximately 42 months)
Population: * Participants were classified as missing or unevaluable if no post-baseline response assessments were available or all post-baseline response baseline assessments were unevaluable.
  * Responders had to have a CR or PR on two consecutive occasions at least 6 weeks apart.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 131 | 135
Percentage of Participants | 13.7 [8.4 to 20.7] | 7.4 [3.7 to 13.0]

9. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Verbatim description of adverse events will be coded to MedDRA preferred terms and graded according to NCI CTCAE v4.0.
Time Frame: Baseline up to end of study (up to approximately 42 month)
Population: The safety population is defined as participants who received any amount of any component of the study treatments (atezolizumab, or enzalutamide). Participants will be allocated to treatment arms according to the treatment they actually received (i.e., participants randomized to enzalutamide alone who received at least one full or partial dose of atezolizumab will be included in the atezolizumab arm for safety)
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 374 | 376
Percentage of Participants
  Total number of participants with at least one adverse event | 96.8 | 92.3
  Total number of participants with at least one treatment related AE | 78.1 | 51.6

10. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Atezolizumab
Description: Safety visit-Discontinued participants had these visits within approximately 120 days after the last dosing; Study Completion Pre-dose visit-Participants had these visits at the last treatment dosing, samples were taken before the last dosing; Early Discontinuation Pre-dose visit-Participants who discontinued the study had these visits within the 30 days after their last dosing but samples were takes before their last dosing; Study Completion visit-Participants had these visits at their last treatment dosing but samples were taken after their last dosing; Early Discontinuation visit-Participants who discontinued the study had the visits within the 30 days after their last dosing but samples were taken after their last dosing; Unscheduled and Unscheduled Pre-dose Visits- At these visits, participants' samples were collected without dosing event and before dosing dosing at a visit unscheduled per protocol respectively. Enzalutamide Arm had no Atezolizumab dosing.
Time Frame: Pre-infusion (0 hour[hr]) on Day 1 Cycles 1, 2, 3, 4, 8, 12, 16 (Cycle length: 21 days); treatment discontinuation visit, 120 days after last dose (up to approximately 42 months)
Population: PK evaluable population. This population is defined as all randomized participants regardless of whether the assigned study treatment was received. For PK analyses, participants were analyzed according to their randomized treatment assignment. Here, "Number Analyzed" refers to number of participants from whom data was collected and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 377 | 0
microgram/mL
  Cycle 1, Day 1, pre-dose: number analyzed (Participants) | 0 | 0
  Cycle 2, Day 1, pre-dose: number analyzed (Participants) | 297 | 0
  Cycle 2, Day 1, pre-dose | 76.4 (69.4) |
  Cycle 3, Day 1, pre-dose: number analyzed (Participants) | 270 | 0
  Cycle 3, Day 1, pre-dose | 124 (79.5) |
  Cycle 4, Day 1, pre-dose: number analyzed (Participants) | 244 | 0
  Cycle 4, Day 1, pre-dose | 147 (65.1) |
  Cycle 8, Day 1, pre-dose: number analyzed (Participants) | 134 | 0
  Cycle 8, Day 1, pre-dose | 157 (305.9) |
  Cycle 12, Day 1, pre-dose: number analyzed (Participants) | 91 | 0
  Cycle 12, Day 1, pre-dose | 155 (497.4) |
  Cycle 16, Day 1, pre-dose: number analyzed (Participants) | 73 | 0
  Cycle 16, Day 1, pre-dose | 137 (144.9) |
  Safety visit: number analyzed (Participants) | 86 | 0
  Safety visit | 2.69 (1759.3) |
  Study Completion/Early Discontinuation: number analyzed (Participants) | 207 | 0
  Study Completion/Early Discontinuation | 82.3 (1008.1) |
  Study Completion/Early Discontinuation pre-dose: number analyzed (Participants) | 2 | 0
  Study Completion/Early Discontinuation pre-dose | 65.3 (106.9) |
  Unscheduled: number analyzed (Participants) | 1 | 0
  Unscheduled | 50.5 (NA) — There was only 1 patient for Cmin Unscheduled visit, therefore CV% mean cannot be calculated. |
  Unscheduled Predose: number analyzed (Participants) | 4 | 0
  Unscheduled Predose | 32.9 (326.5) |

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Atezolizumab
Description: as for outcome 10
Time Frame: Day Cycle 1 Day 1 0.5 hr post-infusion (infusion duration: 60 minutes [min])
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/mL
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 281 | 0
Microgram/mL | 365 (26.5) |

12. Secondary Outcome: Plasma Concentration of Enzalutamide
Description: as for outcome 10
Time Frame: Predose (0 hr) and 1 hr postdose on Day 1 Cycle 1 and 3 (Cycle length: 21 days); pre-dose (within 1 hr) on Day 1 Cycle 8
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/mL
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 141 | 137
Microgram/mL
  Cycle 1 Day 1 Predose: number analyzed (Participants) | 0 | 0
  Cycle 1 Day 1 1 Hr Post: number analyzed (Participants) | 89 | 85
  Cycle 1 Day 1 1 Hr Post | 1.51 (406.4) | 2.42 (270.6)
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 91 | 71
  Cycle 3 Day 1 Predose | 13.1 (29.0) | 13.8 (20.7)
  Cycle 3 Day 1 1 Hr Post: number analyzed (Participants) | 83 | 57
  Cycle 3 Day 1 1 Hr Post | 14.2 (27.3) | 16.0 (19.8)
  Cycle 8 Day 1 Predose: number analyzed (Participants) | 63 | 67
  Cycle 8 Day 1 Predose | 11.3 (103.7) | 12.6 (30.5)
  Unscheduled Predose: number analyzed (Participants) | 0 | 1
  Unscheduled Predose |  | 10.5 (NA) — There was only one patient at unscheduled predose visit, therefore no Geometric Coefficient of Variation values can be calculated

13. Secondary Outcome: Plasma Concentration of N-Desmethyl Enzalutamide
Description: as for outcome 10
Time Frame: as for outcome 12
Population: PK evaluable population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/mL
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 141 | 137
Microgram/mL
  Cycle 1 Day 1 Predose: number analyzed (Participants) | 0 | 0
  Cycle 1 Day 1 1 Hr Post: number analyzed (Participants) | 89 | 85
  Cycle 1 Day 1 1 Hr Post | 0.02 (NA) — N/A represents data that are not evaluable. Lower Than Reportable data. | 0.03 (NA) — N/A represents data that are not evaluable. Lower Than Reportable data.
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 91 | 71
  Cycle 3 Day 1 Predose | 11.9 (33.1) | 11.9 (28.8)
  Cycle 3 Day 1 1 Hr Post: number analyzed (Participants) | 83 | 57
  Cycle 3 Day 1 1 Hr Post | 10.6 (34.2) | 10.9 (29.8)
  Cycle 8 Day 1 Predose: number analyzed (Participants) | 63 | 67
  Cycle 8 Day 1 Predose | 12.8 (36.8) | 13.1 (32.6)
  Unscheduled Predose: number analyzed (Participants) | 0 | 1
  Unscheduled Predose |  | 13.3 (NA) — There was only one patient at unscheduled predose visit, therefore no Geometric Coefficient of Variation values can be calculated

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: The numbers and proportions of ADA-positive participants and ADA-negative participants at baseline (baseline prevalence) and after baseline (post-baseline incidence) will be summarized by treatment group.
  Enzalutamide Arm has no Atezolizumab dosing therefore no participants to include here for Atezolizumab ADA.
Time Frame: Predose (0 hr) on Day 1 Cycles 1, 2, 3, 4, 8, 12, 16 (Cycle length: 21 days); at atezolizumab discontinuation visit (30 days after last dose); 120 days after last dose of atezolizumab; up to 42 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
Number analyzed (Participants) | 386 | 0
Participants
  With Positive Sample at Baseline: number analyzed (Participants) | 370 | 0
  With Positive Sample at Baseline | 2 |
  Without Positive Sample at Baseline: number analyzed (Participants) | 370 | 0
  Without Positive Sample at Baseline | 368 |
  Participants positive for Treatment Emergent ADA: treatment induced: number analyzed (Participants) | 372 | 0
  Participants positive for Treatment Emergent ADA: treatment induced | 52 |
  Participants positive for Treatment Emergent ADA: treatment enhanced: number analyzed (Participants) | 372 | 0
  Participants positive for Treatment Emergent ADA: treatment enhanced | 0 |
  Participants negative for Treatment Emergent ADA: number analyzed (Participants) | 372 | 0
  Participants negative for Treatment Emergent ADA | 320 |

ADVERSE EVENTS:
Time Frame: From Baseline Up To 4 Years 11 Months. For outcome measures and ADA measurements, the time frame was up to 42 (3 years and 6 months) months. However for Adverse Events, the duration of the timeframe was 4 years 11 month. The study was terminated earlier than the planned date and stopped for the efficacy outcomes. And participants' safety was followed up for longer time period.
Description: 4 participants in Atezolizumab + Enzalutamide Arm and 5 participants in Enzalutamide Arm were excluded from the Safety Evaluated Population as they did not receive the study treatment.
  The Safety Evaluated Population comprised with 750 participants (375 and 375 in both arms respectively).
  759 participants who were randomized are included in the At Risk Population for All Cause Mortality.
Arm/Group | Atezolizumab + Enzalutamide | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 219/379 | 191/380
Serious Adverse Events (participants affected / at risk) | 139/374 | 87/376
Other Adverse Events (participants affected / at risk) | 339/374 | 309/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Enzalutamide (N=374) | Enzalutamide (N=376)
Anaemia (Blood and lymphatic system disorders) | 9 (11) | 11 (15)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4) | 2 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 5 (5) | 2 (2)
Chest pain (General disorders) | 3 (3) | 1 (1)
Complication of device insertion (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (4)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (3) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 2 (7)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 10 (13)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Cranial nerve palsies multiple (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 1 (1)
Haematuria (Renal and urinary disorders) | 7 (13) | 5 (7)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Enzalutamide (N=374) | Enzalutamide (N=376)
Anaemia (Blood and lymphatic system disorders) | 83 (98) | 49 (58)
Hypothyroidism (Endocrine disorders) | 21 (22) | 5 (5)
Constipation (Gastrointestinal disorders) | 78 (88) | 62 (65)
Diarrhoea (Gastrointestinal disorders) | 86 (109) | 41 (51)
Nausea (Gastrointestinal disorders) | 86 (95) | 66 (73)
Vomiting (Gastrointestinal disorders) | 31 (35) | 32 (35)
Asthenia (General disorders) | 82 (99) | 63 (68)
Fatigue (General disorders) | 128 (148) | 103 (116)
Oedema peripheral (General disorders) | 33 (38) | 28 (31)
Pain (General disorders) | 24 (26) | 13 (13)
Pyrexia (General disorders) | 31 (37) | 9 (9)
Nasopharyngitis (Infections and infestations) | 13 (15) | 21 (24)
Urinary tract infection (Infections and infestations) | 20 (24) | 18 (21)
Weight decreased (Investigations) | 51 (54) | 32 (33)
Decreased appetite (Metabolism and nutrition disorders) | 115 (129) | 104 (120)
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 (108) | 64 (94)
Back pain (Musculoskeletal and connective tissue disorders) | 80 (98) | 55 (63)
Bone pain (Musculoskeletal and connective tissue disorders) | 27 (31) | 34 (38)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 21 (25) | 15 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (32) | 39 (46)
Dizziness (Nervous system disorders) | 26 (31) | 21 (27)
Headache (Nervous system disorders) | 31 (34) | 19 (21)
Insomnia (Psychiatric disorders) | 29 (29) | 29 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 17 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 17 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 36 (43) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 51 (59) | 10 (10)
Hot flush (Vascular disorders) | 11 (11) | 21 (23)
Hypertension (Vascular disorders) | 27 (33) | 22 (22)
Upper respiratory tract infection (Infections and infestations) | 19 (21) | 14 (15)
Fall (Injury, poisoning and procedural complications) | 21 (26) | 19 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03016312/Prot_SAP_000.pdf